CLINICAL TRIAL: NCT03914859
Title: HAP-REPRO: IMPACT OF POLYCYCLIC AROMATIC HYDROCARBONS (PAH) ON IN VITRO FECONDATION: PARENTAL CELLS WITH EARLY EMBRYONIC QUALITY.
Brief Title: IMPACT OF POLYCYCLIC AROMATIC HYDROCARBONS (PAH) ON IN VITRO FERTILIZATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-32; 2018-A00364 (Registry Identifier: APHM)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Fertilization in Vitro

STUDY DESIGN:
Intervention Model Description: The groups will be defined according to the urinary level of 1-hydroxypyrene, the most sensitive biomarker for PAH exposure. A threshold of 0.1 μmol / mol of creatinine was determined according to the INRS.
  It corresponds to the 90th percentile value for non-smokers not occupationally and nutritionally exposed. The reference value in the general population is <0.51 μg / g creatinine, and in smokers <0.3 μmol / mol creatinine.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed (Other): Urinary level of 1-hydroxypyrene, the most sensitive biomarker of PAH exposure greater than 0.1 μmol / mol creatinine
  Interventions: Biological: IN VITRO FERTILIZATION
- Not exposed (Other): Urinary level of 1-hydroxypyrene, the most sensitive marker of PAH exposure below 0.1 μmol / mol creatinine
  Interventions: Biological: IN VITRO FERTILIZATION

INTERVENTIONS:
Biological: IN VITRO FERTILIZATION — Using exposure biomarker as a reliable means of evaluating gamete quality to estimate the chances of success in in vitro fertilization.

SUMMARY:
The main objective of this study is to highlight a relationship between exposure to PAHs, genotoxic effect biomarkers on spermatozoa and follicular cells, as well as embryonic quality and embryo implantation rates at a given time. IVF attempt. This study therefore analyzes the possibility of using this exposure biomarker as a reliable means of evaluating the quality of gametes in order to estimate the chances of success in IVF.

DETAILED DESCRIPTION:
Objective assessment of the effect of environmental and occupational factors on fertility is difficult to establish due to the lack of relevant exposure biomarkers for reporting multi-exposures.

The main objective of this study is to highlight a relationship between exposure to PAHs, genotoxic effect biomarkers on spermatozoa and follicular cells, as well as embryonic quality and embryo implantation rates at a given time. IVF attempt. This study therefore analyzes the possibility of using this exposure biomarker as a reliable means of evaluating the quality of gametes in order to estimate the chances of success in IVF.

Subsequently, the results of this study will make it possible to personalize and evaluate the effectiveness of the preventive measures put in place upstream of the MPA route by allowing To identify a relationship between PAH exposure and sperm DNA gamete quality in humans, serum AMH concentration and ovarian response to gonadotropic stimulation for IVF in women.

To highlight a relationship between individual exposures to complex PAH mixtures and infertility.

The methodology based, on the feminine side, on the analysis of follicular cells makes it possible to study cells close to female gametes within the cumulo-oocyte complex, without losing the chance of pregnancy for the couple.

ELIGIBILITY:
Inclusion Criteria:

* Couples whose wife is under 36 and the man under 45 at the time of IVF
* Regular cycles of 27 to 33 days in women
* Management of classical IVF (without the use of micro-sperm injection)
* 1st or 2nd attempt of IVF
* Signature of informed consent by both partners of the couple
* Affiliation to a social security scheme or equivalent for both partners of the couple.

Exclusion Criteria:

* Refusal to participate in the study of one or both members of the couple
* No fluency in French
* History likely to alter the ovarian reserve, endometriosis
* Uterine or systemic antecedents, likely to affect implantation
* Andrological antecedents likely to alter fertilization rates
* History of chemotherapy / radiotherapy
* Positive plasma viral load for HIV, HCV or HBV in the year prior to inclusion in one of the members of the couple

Ages: 36 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
expired CO | 72 hours
  The night before the IVF, a urine sample will be collected from both members of the couple, according to the protocol published by the team Partner 2.
  On the day of the IVF, a measurement of the exhaled CO rate will be carried out by the two members of the couple according to the recommendations of the manufacturer.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance des Hôpitaux de Marseille, Marseille, France